CLINICAL TRIAL: NCT05008120
Title: Gut Microbiota in Major Depressive Disorders With and Without Rapid Eye Movement Behavior Disorder: Tracing a Subtype of Depression With Underlying Neurodegeneration
Brief Title: Gut Microbiota in Major Depressive Disorders With and Without Rapid Eye Movement Behavior Disorder
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Health and Medical Research Fund (Other Government)
Responsible Party: Principal Investigator, Professor Wing Yun Kwok, Professor, Chinese University of Hong Kong
Other Study IDs: HMRF18190221
Record Dates: First submitted 2021-08-05; First posted 2021-08-17 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Gut Microbiota
Keywords: Major depressive; Neurodegeneration
MeSH Terms: conditions — Nerve Degeneration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We will perform 16S ribosomal RNA (rRNA) gene sequencing on the fecal microbiome of all individuals. About 20g of the stool sample will be collected from each subject in a sterile container and transferred to the laboratory as soon as possible after collection. All samples arriving in the laboratory will be placed at -80°C before DNA extraction.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- MDD + RBD: 1. Clinical diagnosis of lifetime major depressive disorder, based on the M.I.N.I.;
  2. RBD diagnosis according to the International classification of sleep disorder (ICSD) 3rd edition, fulfilling both the clinical and video-polysomnography (vPSG) criteria;
  3. Depressive symptoms onset before RBD onset
  Interventions: Other: No intervention
- MDD: 1. Age-and sex-matched with MDD+RBD probands;
  2. Lifetime diagnosis of MDD based on M.I.N.I.;
  3. Without a personal history or a family history of RBD or neurodegenerative diseases (i.e. dementia and PD)
  4. Free of RBD symptoms or other hallmark features of RBD (e.g. REM Sleep Without Atonia, RWSA) by vPSG
  Interventions: Other: No intervention
- Health control: 1. Age-and sex-matched with MDD+RBD subjects;
  2. Free of psychiatric disorders based on M.I.N.I.;
  3. Without a personal history or a family history of RBD or neurodegenerative diseases (i.e. dementia and PD)
  4. Free of RBD symptoms or RWSA by vPSG
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The purpose of this study is to identify the variations in gut microbiota compositions between two subtypes of major depressive disorder.

DETAILED DESCRIPTION:
Objective: To identify the variations in gut microbiota compositions between two subtypes of major depressive disorder (MDD), namely those with and without REM sleep behavior disorder (RBD). To correlate the microbiota composition with depressive severity and prodromal markers of α-synucleinopathy.

Design: Case-control study Setting: Established clinical cohorts consisting of patients with comorbid MDD+RBD and MDD only and a group of sexand age-matched healthy control Participants: Patients with comorbid MDD+RBD (n=55), patients with MDD only (n=55), and healthy control (n=55).

Main outcome measures: The abundance and composition of gut microbiota, severity of depressive symptoms, and prodromal markers of α-synucleinopathy.

ELIGIBILITY:
Inclusion Criteria:

1. Age-and sex-matched with MDD+RBD subjects;
2. Free of psychiatric disorders based on M.I.N.I.;
3. Without a personal history or a family history of RBD or neurodegenerative diseases (i.e. dementia and PD)
4. Free of RBD symptoms or RWSA by vPSG

Exclusion Criteria:

1. Presence of narcolepsy and other neurodegenerative diseases that may give rise to RBD and RWSA;
2. Severe psychiatric illness that could not permit a valid written informed consent or otherwise is not suitable for participating in a study;
3. Use of antibiotics within one month and the use of probiotics within three days prior to sample collection;
4. Pre-existing or post-operation of gastrointestinal diseases (e.g. inflammatory bowel disease, gastrointestinal cancer).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The subjects of the current study would be recruited from our established cohort of patients with MDD (with and without RBD). Three groups of subjects are included in the current study, namely healthy control, patients with MDD only, and patients with MDD+RBD.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Composition of gut microbiota | Day 0
  Colonic fecal bacterial composition across two heterogeneous groups of MDD (with and without RBD) and a group of the sex- and age-matched healthy controls

CONTACTS AND LOCATIONS:
Locations (1):
- Shatin Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
Data will be handled and stored under Department of Psychiatry and PI will be responsible for the safekeeping.